CLINICAL TRIAL: NCT06533917
Title: Spinal Cord Stimulation for Chronic Abdominal Pain Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PM23/157561
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main (Experimental): All participants will undergo a single-stage SCS implantation procedure with 2 leads inserted in the posterior epidural space according to standard clinical practice. For ventral column stimulation SCS electrodes will be placed ventrally at T9/10 for upper abdominal pain and at T10/11 to T11/12 for lower abdominal pain.
  Interventions: Device: Main Group

INTERVENTIONS:
Device: Main Group — Thoracolumbar spine AP, Thoracolumbar spine LAT

SUMMARY:
Chronic abdominal pain is a common disorder that can have significant impact on the lives of patients. Treatment options include medication which can have limited effectiveness, be associated with side effects and may lead to tolerance and dependency. Spinal cord stimulation (SCS) is a minimally invasive, therapeutic option for managing chronic abdominal pain. This involves implanting a device that delivers mild electrical signals to the spinal cord to reduce pain. Conventional SCS has been shown to improve abdominal pain caused by different disorders, but it causes feelings of unpleasant tingling in the tummy area. This feasibility study aims to explore relief from chronic abdominal pain symptoms when using a device that does not cause uncomfortable tingling feelings in the tummy area.

DETAILED DESCRIPTION:
Up to 20 patients with chronic abdominal pain will be recruited to participate in this study. They will attend an initial visit prior to having the device implanted and they will be asked to complete a number of questionnaires. Participants will then attend the hospital to have the device implanted and the treatment settings of the stimulation adjusted. Once the stimulation is started, participants will be continuously monitored for their well-being through a series of in-person visits at the pain clinic on a regular basis. These will happen at 1 week and 3, 6 and 12 months after having the device implanted.

ELIGIBILITY:
Inclusion Criteria:

1. Have been clinically diagnosed with CAP (from inguinal crease to T12 ribs), including diagnoses such as abdominal wall pain, chronic pancreatitis, gastroparesis, gastric dysmotility, irritable bowel syndrome, post-surgical or post-traumatic abdominal pain that is of visceral origin.
2. Have been refractory to conservative therapy for a minimum of 3-months, including assessment of at least 2 different classes of medications and/or an anaesthetic block as clinically appropriate.
3. Minimum baseline pain score of 5 on a VAS scale (0-10) for their visceral pain.
4. Be 18 years of age or older at the time of enrolment.
5. Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician.
6. Be willing and capable of giving informed consent.
7. Be willing and able to comply with study-related requirements, procedures, and visits.

Exclusion Criteria:

1. Female participants of childbearing potential who are pregnant/nursing or plan to become pregnant during the trial.
2. Escalating or changing pain condition within the past month as evidenced by investigator examination.
3. Sphlanchnectomy or radiofrequency treatment within the past 6-months.
4. Currently has an active or had an active implantable device including pacemakers, SCS or intrathecal drug delivery system.
5. In the investigators opinion has an active infection.
6. Participated in another clinical investigation within 30-days.
7. Medical co-morbidities that preclude surgical intervention.
8. Participant is incapable of understanding or responding to the study questionnaires.
9. Participant is incapable of understanding or operating the patient programmer handset.
10. Participant is morbidly obese (BMI ≥ 40 kg/m2).
11. Participant has had a spinal surgical procedure or has spinal pathology that would significantly impede lead implantation at the level planned for implantation.
12. Participant has another persistent painful condition other than persistent refractory visceral pain secondary to chronic abdominal pain.
13. History of alcohol abuse in the last year or IV drug abuse in the last 3-years.
14. No increases of more than 40% from baseline amylase.
15. Have a condition currently requiring or likely to require the use of diathermy.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-06-04 (Estimated); Study Completion 2025-06-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and feasibility of ECAP-controlled closed-loop SCS in treating patients with CAP.treating patients with CAP | 12 MONTHS
  To evaluate the safety and feasibility of ECAP-controlled closed-loop SCS in treating patients with CAP.Visual Analogue Scale (VAS) in the last week.
  • Incidence rates of study related adverse events will be collected and characterized.
• Changes in average pain intensity, in the primary region of pain on the Visual Analogue Scale (VAS) in the last week. | 12 MONTHS
  • Changes in average pain intensity, in the primary region of pain on the Visual Analogue Scale (VAS) in the last week.
• Incidence rates of study related adverse events will be collected and characterized. | 12 MONTHS
  • Incidence rates of study related adverse events will be collected and characterized.

CONTACTS AND LOCATIONS:
Overall Officials: Ganesan Baranidharan, MD, Principal Investigator — LTHT
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom